CLINICAL TRIAL: NCT05360017
Title: A Clinical Trial to Evaluate the Effectiveness and Safety of Single Lower Limb Rehabilitation Training Robot in Lower Limb Motor Function Training of Stroke Patients With Hemiplegia
Brief Title: Effectiveness and Safety of Single Lower Limb Rehabilitation Training Robot in Stroke Patients With Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-230
Record Dates: First submitted 2022-03-31; First posted 2022-05-04 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2021-10

CONDITIONS: Hemiplegia
Keywords: hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, controlled, excellent effect, open trial design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot in lower limb motor function training of stroke patients with hemiplegia (Experimental): Test equipment: litestepper single lower limb rehabilitation training robot
  Device type: Class II medical device
  Interventions: Device: litestepper single lower limb rehabilitation training robot

INTERVENTIONS:
Device: litestepper single lower limb rehabilitation training robot — The experimental group adopts litestepper single lower limb rehabilitation training robot walking training on the basis of routine rehabilitation management of stroke patients with hemiplegia, walking training once a day, 40 ± 5 minutes each time; The control group was treated with routine rehabilitation management of stroke patients with hemiplegia. The trial was an open design. Both researchers and subjects knew the treatment allocation and conducted three evaluations within 21 days to evaluate the effectiveness and safety of litestepper single lower limb rehabilitation training robot in the training of lower limb motor function of stroke patients with hemiplegia.

SUMMARY:
This trial is a multi center, randomized, controlled, excellent effect, open and loading trial design. The subjects are randomly assigned to the experimental group and the control group. The experimental group adopts litestepper single lower limb rehabilitation training robot walking training on the basis of routine rehabilitation management of stroke patients with hemiplegia, walking training once a day, 40 ± 5 minutes each time; The control group was treated with routine rehabilitation management of stroke patients with hemiplegia. The trial was an open design. Both researchers and subjects knew the treatment allocation and conducted three evaluations within 21 days to evaluate the effectiveness and safety of litestepper single lower limb rehabilitation training robot in the training of lower limb motor function of stroke patients with hemiplegia.

DETAILED DESCRIPTION:
By collecting the movement gait information of the patient's healthy side limb, judging the patient's movement intention, analyzing and learning the gait characteristics of the patient's healthy side, so as to drive the movement of the single lower limb rehabilitation training robot and drive the patient's affected side limb to carry out the rehabilitation training suitable for the healthy side limb, which can enable the patient to complete the normal walking process and achieve the purpose of auxiliary rehabilitation. Through long-term walking rehabilitation, patients can gradually recover their normal walking gait.

ELIGIBILITY:
Inclusion Criteria:

* understand the whole process of the experiment, voluntarily participate and sign the informed consent;

  * 18-75 years old for both sexes;

    * Stable vital signs, stable condition, tolerance to low-intensity sitting and standing training;

      ④ Weight ≤ 100kg, height 1.50M ~ 1.90m;

      ⑤ Patients with stroke hemiplegia diagnosed as the first onset, including cerebral infarction and intracerebral hemorrhage, the course of disease is within one month after the onset;

      ⑥ One level of sitting or standing balance, able to wear a single lower limb rehabilitation training robot with the help of medical staff;

      ⑦ The passive range of motion of hip and knee is not significantly limited, and the passive range of ankle can be kept in neutral position.

Exclusion Criteria:

* The range of motion of the joint is severely limited and the walking movement is limited;

  * Skin injury or infection of the lower limb in contact with the robot;

    * History of unstable angina pectoris, severe arrhythmia and other heart diseases;

      ④ History of severe chronic obstructive pulmonary disease;

      ⑤ Other contraindications or complications that may affect walking training;

      ⑥ Pregnant women, women preparing for pregnancy or lactation;

      ⑦ Those who participated in any clinical trial within 1 month before enrollment;

      ⑧ Other circumstances that the researcher believes cannot participate in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
The Berg balance scale | Visit three (Day 21 ± 2 ）
  Berg balance scale .The highest score is 56 points and the lowest score is 0 points. The higher the score, the stronger the balance ability. A score of less than 40 indicates a risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jin, Master, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China